CLINICAL TRIAL: NCT06498947
Title: Factors Influencing Physiological Hyperopia in Children: A Prospective Nested Case-control Study
Brief Title: Factors Influencing Physiological Hyperopia in Children
Status: Recruiting | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YH Jiao
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-01

CONDITIONS: Myopia Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Group A is defined as those whose physiological hyperopia (sphere+1/2 cylinder) of at least - 0.5 diopters(D) in either eye.
  Interventions: Other: This study was observational with no intervention.
- Group B: Group B is defined as whose physiological hyperopia exceeds 95% confidence interval for children of same age (Near Myopia).
  Interventions: Other: This study was observational with no intervention.
- Group C: Group C is defined as whose physiological hyperopia exceeds 90% confidence interval for children of same age.
  Interventions: Other: This study was observational with no intervention.

INTERVENTIONS:
Other: This study was observational with no intervention. — This study was observational with no intervention.

SUMMARY:
The trend of myopia in children and its low age is a major social and public health problem in China. More seriously, retinopathy associated with high myopia has become the number one cause of irreversible blinding eye disease in adults in some parts of China. Physiological hyperopia has a protective effect on preventing the onset of myopia, and is one of the strongest predictors of myopia on its own, which is significant in curbing myopia from occurring at a younger age and preventing the development of high myopia before adulthood. However, it is not yet known how the physiological hyperopia changes in childhood, the stage at which the critical inflection point occurs, which key factors lead to the rapid fading of the physiological hyperopia and progression to myopia, and the strength of its effect. In the early stage of the study, the research group established a prospective cohort of preschoolers based on natural population sampling, which included a total of 2109 preschoolers aged 3-6 years from 22 kindergartens in a district in Beijing, and completed a 2-year follow-up, obtaining exploratory results on the changing pattern of physiological hyperopia and key influencing factors in younger children. The group will add new samples to the existing whole cohort sampling cohort and adopt the design scheme of prospective nested case-control study to determine the changing trend of fading trajectory of physiological hyperopia in school-age children, key inflection points and key risk factors, so as to provide new techniques for the prevention and control of childhood myopia.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-9 years old, male or female;
2. Good cooperation in examination;
3. Parents cooperate and sign the informed consent form;

Exclusion Criteria:

1. Children with a history of drug allergy;
2. Pediatric patients with heart disease, cranial trauma or epilepsy, Down syndrome, or glaucoma will be excluded from the cohort.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The research group has already sampled 3-6 years old preschool children from 22 kindergartens in Haidian District, Beijing, and included them in the baseline cohort, which has been followed up continuously for 3 years. The research group will continue to add new samples to the existing cluster sampling cohort and reorganize the cohort of children aged 6-9 years old to conduct this study.
Sampling Method: Probability Sample
Enrollment: 1006 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
myopia | 1 year
  Myopia in this study was defined as an equivalent spherical lens degree ( SER ) error (sphere+1/2 cylinder) of at least - 0.5 diopters(D) in either eye.

SECONDARY OUTCOMES:
Myopia Prevalence | 3 year
  Myopia is defined as a spherical equivalent refractive (SER) (sphere + 1/2 cylinder) of at least -0.5 diopter (D) in either eye.
The change in ocular axis length | 3 year
  The change in ocular axis length was calculated by subtracting each year's measurement from the previous year's measurement.
The change in anterior chamber depth | 3 year
  Calculate the change in anterior chamber depth by subtracting each year's measurement from the previous year's measurement.
The change in corneal curvature | 3 year
  Calculate the change in corneal curvature by subtracting each year's measurement from the previous year's measurement.
The change in the ratio of axial length to corneal curvature | 3 year
  Calculate the change in the ratio of axial length to corneal curvature by subtracting each year's measurement from the previous year's measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Wang J, Li Y, Musch DC, Wei N, Qi X, Ding G, Li X, Li J, Song L, Zhang Y, Ning Y, Zeng X, Hua N, Li S, Qian X. Progression of Myopia in School-Aged Children After COVID-19 Home Confinement. JAMA Ophthalmol. 2021 Mar 1;139(3):293-300. doi: 10.1001/jamaophthalmol.2020.6239. PMID 33443542
- [Result] Saxena R, Vashist P, Tandon R, Pandey RM, Bhardawaj A, Menon V, Mani K. Prevalence of myopia and its risk factors in urban school children in Delhi: the North India Myopia Study (NIM Study). PLoS One. 2015 Feb 26;10(2):e0117349. doi: 10.1371/journal.pone.0117349. eCollection 2015. PMID 25719391
- [Result] He M, Xiang F, Zeng Y, Mai J, Chen Q, Zhang J, Smith W, Rose K, Morgan IG. Effect of Time Spent Outdoors at School on the Development of Myopia Among Children in China: A Randomized Clinical Trial. JAMA. 2015 Sep 15;314(11):1142-8. doi: 10.1001/jama.2015.10803. PMID 26372583
- [Result] Saw SM, Tong L, Chua WH, Chia KS, Koh D, Tan DT, Katz J. Incidence and progression of myopia in Singaporean school children. Invest Ophthalmol Vis Sci. 2005 Jan;46(1):51-7. doi: 10.1167/iovs.04-0565. PMID 15623754
- [Result] Thomson K, Game J, Karouta C, Morgan IG, Ashby R. Correlation between small-scale methylation changes and gene expression during the development of myopia. FASEB J. 2022 Jan;36(1):e22129. doi: 10.1096/fj.202101487R. PMID 34958689
- [Result] Hysi PG, Choquet H, Khawaja AP, Wojciechowski R, Tedja MS, Yin J, Simcoe MJ, Patasova K, Mahroo OA, Thai KK, Cumberland PM, Melles RB, Verhoeven VJM, Vitart V, Segre A, Stone RA, Wareham N, Hewitt AW, Mackey DA, Klaver CCW, MacGregor S; Consortium for Refractive Error and Myopia; Khaw PT, Foster PJ; UK Eye and Vision Consortium; Guggenheim JA; 23andMe Inc.; Rahi JS, Jorgenson E, Hammond CJ. Meta-analysis of 542,934 subjects of European ancestry identifies new genes and mechanisms predisposing to refractive error and myopia. Nat Genet. 2020 Apr;52(4):401-407. doi: 10.1038/s41588-020-0599-0. Epub 2020 Mar 30. PMID 32231278
- [Result] O'Donoghue L, Kapetanankis VV, McClelland JF, Logan NS, Owen CG, Saunders KJ, Rudnicka AR. Risk Factors for Childhood Myopia: Findings From the NICER Study. Invest Ophthalmol Vis Sci. 2015 Feb 5;56(3):1524-30. doi: 10.1167/iovs.14-15549. PMID 25655799
- [Result] Flitcroft DI, He M, Jonas JB, Jong M, Naidoo K, Ohno-Matsui K, Rahi J, Resnikoff S, Vitale S, Yannuzzi L. IMI - Defining and Classifying Myopia: A Proposed Set of Standards for Clinical and Epidemiologic Studies. Invest Ophthalmol Vis Sci. 2019 Feb 28;60(3):M20-M30. doi: 10.1167/iovs.18-25957. PMID 30817826
- [Result] Zadnik K, Sinnott LT, Cotter SA, Jones-Jordan LA, Kleinstein RN, Manny RE, Twelker JD, Mutti DO; Collaborative Longitudinal Evaluation of Ethnicity and Refractive Error (CLEERE) Study Group. Prediction of Juvenile-Onset Myopia. JAMA Ophthalmol. 2015 Jun;133(6):683-9. doi: 10.1001/jamaophthalmol.2015.0471. PMID 25837970
- [Result] Matsumura H, Hirai H. Prevalence of myopia and refractive changes in students from 3 to 17 years of age. Surv Ophthalmol. 1999 Oct;44 Suppl 1:S109-115. doi: 10.1016/s0039-6257(99)00094-6. PMID 10548123
- [Result] French AN, Morgan IG, Mitchell P, Rose KA. Risk factors for incident myopia in Australian schoolchildren: the Sydney adolescent vascular and eye study. Ophthalmology. 2013 Oct;120(10):2100-8. doi: 10.1016/j.ophtha.2013.02.035. Epub 2013 May 11. PMID 23672971
- [Result] Morgan IG, French AN, Ashby RS, Guo X, Ding X, He M, Rose KA. The epidemics of myopia: Aetiology and prevention. Prog Retin Eye Res. 2018 Jan;62:134-149. doi: 10.1016/j.preteyeres.2017.09.004. Epub 2017 Sep 23. PMID 28951126
- [Result] Cui Y, Zhang L, Zhang M, Yang X, Zhang L, Kuang J, Zhang G, Liu Q, Guo H, Meng Q. Prevalence and causes of low vision and blindness in a Chinese population with type 2 diabetes: the Dongguan Eye Study. Sci Rep. 2017 Sep 11;7(1):11195. doi: 10.1038/s41598-017-11365-z. PMID 28894238
- [Result] Iwase A, Araie M, Tomidokoro A, Yamamoto T, Shimizu H, Kitazawa Y; Tajimi Study Group. Prevalence and causes of low vision and blindness in a Japanese adult population: the Tajimi Study. Ophthalmology. 2006 Aug;113(8):1354-62. doi: 10.1016/j.ophtha.2006.04.022. PMID 16877074
- [Result] Wong TY, Ferreira A, Hughes R, Carter G, Mitchell P. Epidemiology and disease burden of pathologic myopia and myopic choroidal neovascularization: an evidence-based systematic review. Am J Ophthalmol. 2014 Jan;157(1):9-25.e12. doi: 10.1016/j.ajo.2013.08.010. Epub 2013 Oct 5. PMID 24099276
- [Result] Li SM, Liu LR, Li SY, Ji YZ, Fu J, Wang Y, Li H, Zhu BD, Yang Z, Li L, Chen W, Kang MT, Zhang FJ, Zhan SY, Wang NL, Mitchell P; Anyang Childhood Eye Study Group. Design, methodology and baseline data of a school-based cohort study in Central China: the Anyang Childhood Eye Study. Ophthalmic Epidemiol. 2013 Dec;20(6):348-59. doi: 10.3109/09286586.2013.842596. Epub 2013 Oct 25. PMID 24160405